CLINICAL TRIAL: NCT03384771
Title: Predictors of Outcomes in MBSR Participants From Teacher Factors
Acronym: Prompt-F
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Massachusetts, Worcester (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R34AT008948 (NIH); 1R34AT008948 (NIH)
Record Dates: First submitted 2017-06-11; First posted 2017-12-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: mindfulness, MBSR, teaching
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MBSR Students: community-dwelling adults who register for relevant MBSR courses at University of Massachusetts Center for Mindfulness (UMass CFM), University of California San Francisco (UCSF), or participating community sites
  Interventions: Behavioral: MBSR
- MBSR Teachers: those teaching MBSR courses at UMass CFM, UCSF, or participating community sites
- Raters: experience mindfulness teachers, recruited by invitation, who will participate in MBI-TAC training

INTERVENTIONS:
Behavioral: MBSR — There is no study intervention per se, but participants will be teaching or enrolled in public 8-week MBSR classes.
  Other Names: Mindfulness Based Stress Reduction
  Groups: MBSR Students

SUMMARY:
Objectives. The primary objective of the current proposal is to identify teacher-related factors that can be feasibly measured and shown to predict mindfulness-based intervention (MBI) participant outcomes. The secondary objective of this R34 proposal is to lay the groundwork for a large-scale R01-funded study in which the investigators anticipate studying participants in Mindfulness-Based Stress reduction (MBSR) courses provided by 50 or more teachers in a range of university- and community-based settings.

DETAILED DESCRIPTION:
Objectives. The primary objective of the current proposal is to identify teacher-related factors that can be feasibly measured and shown to predict mindfulness-based intervention (MBI) participant outcomes. The secondary objective of this R34 proposal is to lay the groundwork for a large-scale R01-funded study in which the investigators anticipate studying participants in Mindfulness-Based Stress reduction (MBSR) courses provided by 50 or more teachers in a range of university- and community-based settings. Design and Outcomes. This is an observational study of MBSR participants, teachers, and raters. Student participants will receive recruitment videos of different lengths and varying compensation schedules; The study will examine these to optimize participation and retention in the future R01 study.

Interventions and Duration. There is no study intervention per se, but participants will be teaching or enrolled in public 8-week MBSR classes. Outcome data will be collected from participants using internet-administered questionnaires at baseline, 2 months (immediate post-MBSR) and 4 months (post-MBSR follow-up). Rater study: The investigators will invite experience meditation teachers to be trained to use a the Mindfulness-Based Interventions Teaching Assessment Criteria (MBI-TAC) tool as a standardized approach to rating MBSR teacher competency. As part of the training, the study will be collecting data on how the training works. Thus, those who join the training will be asked to sign a consent form and complete a brief questionnaire about their teaching and meditation experience, as well as demographics; the study will also collect data on the ratings they do as part of the training. The goal of this part of the study is to assess the rater-training process.

Sample Size and Population. The study aims to enroll about 19 MBSR teachers and 200 MBSR participants, along with about 30 raters to be trained in the MBI-TAC system.

ELIGIBILITY:
Teachers

Inclusion Criteria:

* teaching MBSR in one of the study recruitment sites during the study period
* choose to participate

Exclusion:

• none

MBSR Participants

Inclusion Criteria:

* enrolled in MBSR class taught by an enrolled teacher
* choose to participate
* age 18 years or older

Exclusion:

• none

Raters

Inclusion Criteria:

* Certified to teach MBSR through the CFM's OASIS (or equivalent) training program.
* 3+ years of MBSR teaching experience, having taught 10 MBSR classes.
* 10+ years of personal mindfulness practice with daily practice and yearly retreat experience (on average 5+ days).
* Have the interest and time available to complete web-based rater training and subsequent teacher ratings using an online interface, including in the Testing Phase.
* Ideally will be able to attend at least 7/8 training dates.

Exclusion:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MBSR Teachers MBSR Participants MBI-TAC Raters
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
MBI-TAC inter-observer variability | 2 months
  The key metric to be used to evaluate inter-observer variability is intraclass-correlation (ICC). 1 ICC provides a measure of how strongly ratings of the same item by different raters resemble each other, with values ranging from 0 (only random agreement) to 1 (perfect agreement). ICC will be calculated for each of the six domains in MBI:TAC, as well as the summary score.

SECONDARY OUTCOMES:
Rater agreement | 4 months
  Rater agreement
Rater test-retest reliability | 4 months
  Rater test-retest reliability
Distinguishing novice from experienced MBSR teachers | 2 months
  The difference in ratings of novice and experienced teachers with raters blinded to teacher experience will be examined. Comparison of mean scores will be performed using t-tests to compare mean scores between dichotomously grouped teachers (novice vs. experienced), and regression to test associations with ratings using experience as an ordinal variable (by grouped years of experience).
Participant rating of teachers | 2 months
  Internal consistency of the multiple items meant to measure each domain of teacher quality (e.g. coverage and pacing) using Cronbach's alpha. Scores on questions for each domain will be averaged to provide an overall score for the domain. ICC will be tested for each domain in a similar fashion to that described for the MBI:TAC; note that lower ICC values are anticipated on this instrument than the MBI:TAC, given the varied perspectives of different participants. Finally, the correlation of participant ratings of each domain (averaging ratings across participants) to ratings from the MBI:TAC.blinded to teacher experience will be tested. Comparison of mean scores will be performed using t-tests to compare mean scores between dichotomously grouped teachers (novice vs. experienced), and regression to test associations with ratings using experience as an ordinal variable (by grouped years of experience).
Patient Reported Outcome Measurement Information System (PROMIS-29) Fatigue scale | 2 months
  Higher scores indicate more fatigue (worse outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Patient Reported Outcome Measurement Information System (PROMIS-29) Depression scale | 2 months
  Higher scores indicate more depression (worse outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Patient Reported Outcome Measurement Information System (PROMIS-29) Sleep Disturbance scale | 2 months
  Higher scores indicate more Sleep Disturbance (worse outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Patient Reported Outcome Measurement Information System (PROMIS-29) Physical Function scale | 2 months
  Higher scores indicate more Physical Function (better outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Patient Reported Outcome Measurement Information System (PROMIS-29) Pain Interference scale | 2 months
  Higher scores indicate more Pain Interference (worse outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Patient Reported Outcome Measurement Information System (PROMIS-29) Pain Intensity scale | 2 months
  Higher scores indicate more Pain Intensity (worse outcome). PROMIS-29 scales use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric, a score of 40 is one SD lower than the mean of the reference population, while score of 60 is one SD higher than the mean of the reference population. Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Perceived Stress Scale-short | 2 months
  Stress appraisal, 4 items. Range: 0-16, higher scores indicate greater perceived stress (worse outcome).
Five Facet Mindfulness Questionnaire-short form (FFMQ-SF) | 2 months
  Mindfulness in five domains: observing, describing, acting with awareness, not judging inner experience, and not reacting to inner experience, 24 items Total score Range: 24-120, with higher scores indicating greater mindfulness (better outcome).
  Subscale Ranges: For describe, act with awareness, and non-judge, and non-react (all 5-item subscale): 5-25. For observe (4-items): 4-20. Higher scores indicate greater mindfulness (better outcome).
Positive Affect from the Positive and Negative Affect Scale (PANAS) | 2 months
  Intensity of positive emotions, 10 items.Range: 10-50, higher scores represent higher levels of positive affect (better outcome)
Negative Affect from the Positive and Negative Affect Scale (PANAS) | 2 months
  Intensity of negative emotions, 10 items. Range: 10-50, higher scores represent higher levels of negative affect (worse outcome)
Self-Compassion Scale (SCS-SF) | 2 months
  12 items. Range: 12-60, higher scores indicate greater self-compassion (better outcome).
Expected and Perceived benefit of MBSR | 2 months
  Participant expectations of and perceived benefit of the MBSR course, 5 items--Benefit overall, handling stress, managing mood/emotions, relationships, and physical health problems. Items can be summed to create total benefit score. Range: 0-50, with higher scores indicating greater benefits. Range for the individual items: 0-10, with higher scores indicating greater benefits (better outcome).
Study retention | 2 months
  Effects of video length and compensation factors on student retention in the study
Study enrollment | 0 months
  Effects of video length and compensation factors on enrollment into the study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Osher Center for Integrative Medicine, San Francisco, California
  - Center for Mindfulness at University of Massachussets, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided